CLINICAL TRIAL: NCT03669432
Title: Phase II Randomized Controlled Trial Of Postoperative Intensity Modulated Radiotherapy (IMRT) in Locally Advanced Thyroid Cancers.
Brief Title: To Study the Impact of Radiation Treatment After Surgery in Patient With Locally Advanced Thyroid Cancer.
Acronym: THYRO-RT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Department of Atomic Energy (Other Government)
Responsible Party: Principal Investigator, Dr. Gouri Pantvaidya, Associate Professor & Assistant surgeon E, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1076
Record Dates: First submitted 2018-05-04; First posted 2018-09-13 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Thyroid Cancer Stage IV; Radiation Toxicity
Keywords: locally advanced thyroid cancers, IMRT, toxicity
MeSH Terms: conditions — Thyroid Neoplasms; Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensity Modulated radiotherapy (Experimental): In this Arm, after surgery, patient will receive radio-iodine treatment as per guidelines, 6-8 weeks after surgery. The patient will receive adjuvant radiation therapy about 8-10 weeks after completion of initial surgery. The duration of this radiation therapy will be approximately 45 days.
  : The goal of the treatment plan would be to encompass the PTV subclinical disease with a dose of 54-60 Gy and the PTV of the gross disease with 70-74 Gy while sparing as much of the aforesaid critical structures as possible.
  The maximum permissible point doses to the spinal cord will be limited to 46 Gy. IMRT planning and delivery will be carried out on the Tomotherapy Hi Art System.
  Interventions: Radiation: Intensity Modulated Radiotherapy; Procedure: Surgery alone
- Surgery alone (Other): In this Arm, after surgery patient will receive radio-iodine treatment as per guidelines, 6-8 weeks after surgery. Patient under surgery arm will receive no further treatment after surgery and radio-iodine therapy and will be kept on a routine follow up
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy — The patient will receive adjuvant radiation therapy about 8-10 weeks after completion of initial surgery. The duration of this radiation therapy will be approximately 45 days.
  : The goal of the treatment plan would be to encompass the PTV subclinical disease with a dose of 54-60 Gy and the planned target volume (PTV) of the gross disease with 70-74 Gy while sparing as much of the aforesaid critical structures as possible.
  The maximum permissible point doses to the spinal cord will be limited to 46 Gy. IMRT planning and delivery will be carried out on the Tomotherapy Hi Art System.
  Arms: Intensity Modulated radiotherapy
Procedure: Surgery alone — This intervention is of no interest

SUMMARY:
This trial deals with cancers of the thyroid gland which are advanced at the local site of thyroid. These cancers are treated with surgery and complete removal of the thyroid gland. But due to advanced nature, there is risk of re-occurrence. Radiotherapy can be used to prevent this re-occurrence. This study attempt to see the effect of radiotherapy in preventing re-occurrence and its side effects in advanced thyroid cancer.

DETAILED DESCRIPTION:
Surgery, when possible offers the best chance of cure for cancer of the thyroid gland. Surgery for thyroid cancer involves removal of the thyroid gland along with removal of the lymph nodes which drain the gland. After surgery most patients will receive radio-iodine treatment to diagnose and treat any spread of the cancer in the body. Most thyroid cancers will have good outcomes with the above mentioned treatment. However, in advanced thyroid cancer there is a higher chance of recurrence even with surgery and radio iodine. Surgery for recurrence of these cancers is very morbid This may entail surgeries which may also involve removing portions of the voice box and food pipe. You may therefore develop and discomfort or inability to eat or speak.

Radiation therapy can be given to the neck along with radio-iodine therapy to decrease these re occurrences of the cancer. A number of studies have shown a benefit with the use of radiation therapy in advanced cases of thyroid cancer. However, the side effects of radiation, if any, have not been well documented. This study is being done to assess the impact of radiation on the outcome of cancer and the exact side effects of radiation therapy. If the side effects are not too many, then radiation therapy can be used to decrease the chances of recurrence in the neck after thyroid.

In this study, patients undergoing total thyroidectomy for thyroid cancer will be assessed for high risk features on the histopathology report and the intra operative findings. Those with advanced thyroid cancer as per the eligibility criteria will be counselled and consented for the study. Those patients willing to participate in the study will be randomised to either receive only surgery and radio-iodine or surgery, radio-iodine and external beam radiation.

ELIGIBILITY:
Inclusion Criteria:

A) All patients of differentiated thyroid cancer (papillary/follicular/poorly differentiated/) who have undergone total/completion thyroidectomy at our institute and having at least two of the following features (listed below) intra-operatively and/or on histopathology

1. Gross extrathyroidal spread into soft tissues of the neck, trachea, esophagus, recurrent laryngeal nerve (constituting stage T4a)
2. R1/ shave resections (minimal residual disease)
3. R2 resections (gross residual disease)
4. Multiple lymph nodes positive(>2) with perinodal extension at level VI B) Normal baseline haematological and biochemical parameters.

Exclusion Criteria:

1. Anaplastic or medullary thyroid cancer
2. Previous history of radiation
3. Pregnancy
4. < 18 years Patient unwilling to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
locoregional recurrence | after completion of treatment- till 5 years
  locoregional recurrence is defined as occurrence of pathology proven recurrence in the neck

SECONDARY OUTCOMES:
acute toxicity | during treatment- till 23 months
  Acute toxicity will be measured during and after completion of radiation (3 months).
late toxicity | at 2 years after treatment completion
  Late toxicity will be measured using the LENT-SOMA scale

CONTACTS AND LOCATIONS:
Locations (1):
- Gouri Pantvaidya, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT03669432/Prot_SAP_001.pdf
  • Informed Consent Form (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03669432/ICF_000.pdf